CLINICAL TRIAL: NCT00000802
Title: A Randomized, Comparative Study of Daily Dapsone and Daily Atovaquone for Prophylaxis Against PCP in HIV-Infected Patients Who Are Intolerant of Trimethoprim and/or Sulfonamides
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 277; CPCRA 034; 11253 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Dapsone; Antifungal Agents; Acquired Immunodeficiency Syndrome; atovaquone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atovaquone; Dapsone

INTERVENTIONS:
Drug: Atovaquone
Drug: Dapsone

SUMMARY:
To compare the efficacy and safety of dapsone versus atovaquone in preventing or delaying the onset of histologically proven or probable Pneumocystis carinii pneumonia in HIV-infected patients with CD4 counts <= 200 cells/mm3 or <= 15 percent of the total lymphocyte count who are intolerant to trimethoprim and/or sulfonamides.

Trimethoprim/sulfamethoxazole (TMP/SMX), which is effective for secondary PCP prophylaxis, is associated with allergic manifestations and side effects that limit its use. Patients who are intolerant of TMP/SMX require an effective alternative. Dapsone and atovaquone have both shown promise as PCP prophylactic agents.

DETAILED DESCRIPTION:
Trimethoprim/sulfamethoxazole (TMP/SMX), which is effective for secondary PCP prophylaxis, is associated with allergic manifestations and side effects that limit its use. Patients who are intolerant of TMP/SMX require an effective alternative. Dapsone and atovaquone have both shown promise as PCP prophylactic agents.

Patients are randomized to receive either dapsone or atovaquone daily, with follow-up at the clinic every 4 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Strongly recommended:

* Pyrimethamine (50 mg) and folinic acid (15 mg) weekly in patients receiving dapsone who have CD4 count < 100 cells/mm3 and are toxoplasmosis seropositive.

Patients must have:

* Working diagnosis of HIV infection.
* CD4 count <= 200 cells/mm3 or <= 15 percent of total lymphocyte count at any time in the past OR a history of PCP.
* History of intolerance of trimethoprim and/or sulfonamides that required permanent discontinuation.

NOTE:

* Pregnant patients are eligible at the clinician's discretion.

Prior Medication:

Allowed:

* Prior PCP prophylaxis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active pneumocystosis.

Concurrent Medication:

Excluded:

* PCP prophylaxis (other than study drug) or any medication with potential anti-PCP activity.

Patients with the following prior conditions are excluded:

* Known treatment-limiting reaction to dapsone or atovaquone.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Study Completion 1997-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: El-Sadr W, Study Chair; Luskin-Hawk R, Study Chair; Murphy R, Study Chair
Locations (44):
- United States (43):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Emory Univ. Hemophilia Program Office, Atlanta, Georgia
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Wake County Health and Human Services CRS, Raleigh, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] El-Sadr WM, Murphy RL, Yurik TM, Luskin-Hawk R, Cheung TW, Balfour HH Jr, Eng R, Hooton TM, Kerkering TM, Schutz M, van der Horst C, Hafner R. Atovaquone compared with dapsone for the prevention of Pneumocystis carinii pneumonia in patients with HIV infection who cannot tolerate trimethoprim, sulfonamides, or both. Community Program for Clinical Research on AIDS and the AIDS Clinical Trials Group. N Engl J Med. 1998 Dec 24;339(26):1889-95. doi: 10.1056/NEJM199812243392604. PMID 9862944
- [Background] Caldwell P, Murphy R, Chan C, Yurik T, Scott J, el-Sadr W. Atovaquone suspension (ATQ) for prophylaxis of Pneumocystis carinii pneumonia (PCP): effects of baseline prophylaxis on safety and efficacy. Int Conf AIDS. 1998;12:297 (abstract no 22178)
- [Background] Murphy R, El-Sadr W, Cheung T, Luskin-Hawk R, Yurik T, Neaton J, Hafner R. Impact of protease inhibitor containing regimens on the risk of developing opportunistic infections and mortality in the CPCRA 034/ACTG 277 study. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:113 (abstract no 181)